CLINICAL TRIAL: NCT03810326
Title: Safety and Efficacy of a Device for the Relief of Pain Due to Carpal Tunnel Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yuinvent Innovations Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VY-CTS1-01
Record Dates: First submitted 2019-01-17; First posted 2019-01-18 (Actual); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental)
  Interventions: Device: CTR device (tradename named Xtend)

INTERVENTIONS:
Device: CTR device (tradename named Xtend) — Non invasive active splint

SUMMARY:
Interventional study to evaluate efficacy and safety of an active splint.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, above 40 years of age.
* Able to understand and sign informed consent
* Pain associated with mild to moderate carpal tunnel syndrome in a single wrist
* Numbness and tingling in the median nerve distribution
* Nocturnal Numbness
* Weakness and/or atrophy of the thenar musculature
* Demonstrate positive Phalen's Test of the affected extremity
* Demonstrate positive Tinel's Test of the affected extremity
* Sensory impairment defined as a loss of 2-point discrimination
* Have recent (within 3 months) electro-diagnostic evidence of Carpal Tunnel Syndrome

Exclusion Criteria:• Currently receiving treatment for carpal tunnel syndrome

* History of surgical carpal tunnel release
* Pregnancy
* Diabetes not controlled by medication
* Radiculopathy i.e., cervical radiculopathy, diabetic radiculopathy
* Thoracic outlet syndrome
* Compromised skin integrity
* Past history of traumatic event, surgery, or congenital impairment of the forearm, wrist, or hand

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-01-12 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
Reduction in pain score | 10 weeks
  Reduction in NRS reported pain score

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No